CLINICAL TRIAL: NCT06351839
Title: Metacognitive Behavioral Therapy Integrated in Sleep Treatment for Comorbid Insomnia in Patients With Persistent Pain: A Randomized Controlled Semi-Crossover Clinical Trial
Brief Title: Sleep Well Despite Persistent Pain Symptoms
Acronym: Sleep-Well
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tromso (Other)
Collaborators: University Hospital of North Norway (Other); Diakonhjemmet Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2024/500457(REK)
Record Dates: First submitted 2024-02-29; First posted 2024-04-08 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2024-03

CONDITIONS: Insomnia Chronic; Insomnia Due to Medical Condition; Pain, Chronic
Keywords: Insomnia; Comorbid insomnia; Chronic pain; MetaCognitive Therapy for Insomnia; Sleep Hygiene; Sleep Education; Sleep Restriction; Group therapy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Chronic Pain; Sleep Hygiene

STUDY DESIGN:
Intervention Model Description: We randomize patients to receive either the Sleep-Well intervention or to the TAU condition (active waiting-list group). After 3 months, the TAU patients cross over and receive the Sleep-Well intervention; hence, the design is semi-crossover.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TAU control arm (Active Comparator): The treatment-as-usual arm.
  Interventions: Behavioral: TAU (treatment-as-usual)
- The Sleep-Well intervention (Experimental): The study arm that receives the Sleep-Well intervention.
  Interventions: Behavioral: Sleep-Well despite persistent pain

INTERVENTIONS:
Behavioral: Sleep-Well despite persistent pain — The Sleep-Well program covers four overarching topics stretched over 7 group sessions (each lasting ~1.5 hours): 1) providing information about sleep physiology, causes of sleep problems, sleep habits and hygiene and use of sleep assessment methods (i.e., sleep diaries) for deciding sleep restriction schedules; 2) behavioural strategies through the application of stimulus control and sleep restriction; , 3) mental strategies by addressing and changing unhelpful (meta)cognitions that commonly occur in sleep and persistent pain conditions; and 4) strategies related to maintenance of good sleep and prevention of relapse. The program has been developed by Diakonhjemmet hospital in Oslo and includes a guideline for therapist and a workbook for patients (that includes home tasks for the participant).
  Arms: The Sleep-Well intervention
Behavioral: TAU (treatment-as-usual) — The treatment-as-usual arm represents an active waiting-list arm as subjects receive standard care, which may involve some sleep assessment, rudimentary advice/education about sleep, and possibly also sleep medication. The type of sleep treatment this group receives during the waiting-list period will be recorded from the patients' journal.
  Arms: TAU control arm

SUMMARY:
Background: The prevalence of comorbid insomnia is 8-10 times higher in patients with chronic pain than in the general population. Insomnia adds a considerable burden as it worsens the quality of life, restoration and repair, mental health and pain symptoms. Since pain and sleep problems are mutually reinforcing, improvements in sleep may have beneficial effects on pain. Unfortunately, the customary use of sleep medication (TAU: treatment-as-usual) often yields short-lived plus side effects. The "Sleep-Well" intervention examines if a group-based intervention program focusing on sleep literacy, sleep restriction, stimulus control and metacognitive therapy modules may perform better than TAU in improving patients' insomnia and sleep quality.

Eligible patients: Investigators target adult patients referred to the University Hospital of North Norway (Tromsø) for a diagnostic evaluation of their pain condition. Patients eligible for the Sleep-Well study are those who satisfy diagnostic criteria for a non-malign pain disorder plus a comorbid insomnia sleep disorder. Patients are not eligible if they use drugs or large doses of morphine (>100 equivalents), are engaged in an insurance case due to their diagnosis, or participate in other ongoing group programs at the hospital.

Aims: This trial uses a randomized semi-crossover design to examine if the Sleep-Well group does better regarding insomnia and sleep quality than the control patients (TAU). The primary outcome measures are reductions in diagnostic criteria for insomnia, self-reported insomnia symptoms, quality of life, and actigraphy-measured insomnia indicators (long sleep onset latency, frequent nightly awakenings and early morning awakening). The secondary outcome measures include a simplified polysomnography measurement of brain activity during sleep to assess if proportions or durations of slow-wave versus light-wave sleep and EEG-based arousal indices improve. In addition, it is examined if the Sleep-Well intervention incurs benefits concerning pain complaints, dysfunctional sleep and pain cognitions, anxiety and depression.

The intervention: The Sleep-Well program schedules group sessions that cover four topics (sleep literacy, behavioural and mental strategies, maintenance and relapse prevention). All sessions are led by two therapists. Those randomized to the active control group (TAU) cross over to the Sleep-Well intervention three months later.

DETAILED DESCRIPTION:
Background: Insomnia is 8-10 times more prevalent among patients with chronic pain than in the general population. The disrupted sleep restoration caused by insomnia can be exhausting for the patient as insomnia also impairs pain inhibition. Sleep medications often yield short-lived clinical responses and further introduce risks of "hangover", tolerance, and even addiction. Psychological sleep treatment is thus clearly preferable given sufficient effect.

Cognitive Behavioral Therapy is the recommended first-line treatment of insomnia (CBT-i). Psychological interventions are also recognized in the treatment and follow-up of chronic pain. However, the evidence of psychological treatment of comorbid insomnia in patients with chronic pain is very limited, although some few results are promising .

Insomnia is the most common sleep disorder and involves nocturnal symptoms (e.g. long sleep onset latency, nightly awakenings, and early morning awakening) and daytime problems (e.g. fatigue, mood swings, concentration difficulties, impaired function at work, school, or in social life). Acute insomnia symptoms triggered by adverse life events or acute illnesses are normal, whereas the transition to chronic insomnia is not. Chronic pain is a chronic stressor and may act both as a precipitating and perpetuating factor for insomnia, generating high levels of stress-activating hormones.

Rumination on the causes of pain is frequently observed in chronic pain, often combined with a cognitive inclination towards catastrophizing (i.e., repetitive, intrusive, and difficult-to-ignore thoughts). Meta-cognitions, such as rumination and catastrophizing may perpetuate insomnia by maintaining a high level of sleep-disruptive psychophysiological arousal and loss of deep sleep. Affective and anxiety disorders are other frequent comorbidities of chronic pain, that may further aggravate the effects of rumination and catastrophizing on both sleep and pain.

Meta-Cognitive Therapy (MCT) has well-documented effects on depression and anxiety disorders. Studies of MCT in insomnia are limited, which is unfortunate as it seems to modulate symptoms substantially across multiple health conditions. The advantage of MCT is the focus on how one relates to, evaluates, monitors, or reacts emotionally to internal thoughts rather than their specific content or experienced truth as in CBT. Change in dysfunctional cognitions about sleep is a central element of CBT-i. The strong association between insomnia and sleep-related metacognitions (thought patterns), rather than negative sleep-related cognitions (thought content), suggests that psychological treatment of insomnia should include MCT.

The sleep intervention for the present intervention study (hereafter "Sleep-Well") applies a modified version of a Norwegian CBT-i manual by the Diakonhjemmet hospital in Oslo, integrating elements of MCT. Sleep-Well is group-based and covers four modules; i.e. 1 (introduction), information about sleep physiology, causes of sleep problems, sleep hygiene and the use of sleep diaries; 2 (behavioral strategies), concerns stimulus control and sleep restriction; 3 (cognitive strategies) represent a CBT/MCT part focusing on sleep-disturbing cognitions and metacognition common to pain and sleep; and 4, maintenance and prevention of relapse.

Hypotheses: This trial examines if the Sleep-Well intervention performs better than the "treatment as usual" (TAU) group, i.e., rudimentary sleep evaluation and education plus sleep medication on indication, in terms of statistically significant improvements in:

1. (primary hypotheses) self-reported insomnia symptoms, diagnostic criteria for insomnia, health-related quality of life, and actigraphy recorded indicators of insomnia (i.e., SOL-sleep onset latency, WASO-wakeup after sleep onset, EMA-early morning awakening and SE-sleep efficiency).
2. (secondary hypotheses) self-reported symptoms of fatigue, symptoms of anxiety and depression, pain-symptoms related to acceptance, intensity and interference, and need for sleep medication. In addition, improvements in objective sleep recordings (the Home Sleep Test) related to the proportion and duration of slow-wave sleep periods, and sleep disturbance as indicated by the EEG-based arousal-index.

In addition, this trial explores

* whether mediator variables as described in the Measurement Outcomes section (under other variables) may identify treatment mechanisms related to the Sleep-Well program.
* through qualitative interviews participants' perceived feasibility and acceptability of Sleep-Well, and if qualitative contrasts are present between those benefitting well versus poorly with regard to primary insomnia symptoms.

Study design and procedures: This study uses a randomized semi-crossover design. Participants are randomized to the Sleep-Well or the active treatment-as-usual (TAU) comparator condition receiving standard sleep treatment at the hospital or their general practitioner. Participants are block randomized (block size = 4) to maintain equal treatment and TAU group sizes. After three months of waiting time, the TAU participants cross over to the Sleep-Well group.

The outcome measurements are registered at baseline (before the randomization), and after finishing the Sleep-Well intervention (posttest ~3 months). In addition, we conduct two follow-ups at three and 12 months to examine relapse. The TAU group carries out two pre-tests (before randomization, and before initiation of Sleep-Well) to control for sleep function changes during the waiting period.

Statistical power and analyses Power calculation: A meta-analysis of comparable somatic diagnoses (5 studies) indicated a standardized mean difference (Cohen´s d) between intervention and control ranging between 0.60-0.80 (Tang et al., 2015). With randomization done on an individual level, a correlation = 0.5 between pre- and post-test (R-sq=25%), alpha = 0.05, power = 0.80, and minimum Cohen´s d = 0.60, at least N = 68 patients are required to reject the null hypothesis. With an estimate of ICC (intra-class correlation) = .05 (adjustment for similarities that occur between patients due to sharing of a treatment group, cluster size=6), which yields a design effect of 1.25 (1+(6-1)*ICC), at least N = 85 participants are needed. By adding a safety margin of 20% dropout, the final sample estimate is N = 106 patients.

Statistical analyses: Generalized linear mixed models (GenLinMixed) are used as a general rule due to great flexibility in handling both continuous, binary, and count-based outcome variables, and estimation of random effects for adjustment purposes due to dependency in the outcome measures at different levels (e.g. repeated data, treatment group clusters). The analyses are carried out conservatively as intention-to-treat. Alpha < .05 and .01 are assumed for the hypotheses about primary sleep treatment outcomes (insomnia, sleep quality) and secondary/exploratory treatment effects (affective health, fatigue, quality of life) and moderators/mediators, respectively.

Qualitative analyses: The transcribed semi-structured interview data will be analyzed using the reflexive thematic analysis methodology, which across five steps seeks to identify the number of overall conceptual dimensions that meaningfully account for all the interview texts. The Consolidated Criteria for Reporting Qualitative Research will be applied.

Interaction with user representatives: The project has included two user representatives with first-hand experiences with chronic pain. They actively participate in multiple parts of the research process and are particularly consulted in questions related to relevance (e.g., regarding questionnaires and the content of Sleep-Well), the process of implementing the Sleep-Well intervention, and on issues related to avoiding over-burdening the participants.

Ethics: The Sleep-Well study has been approved by the Regional Committee for Medical and Health Research Ethics (CaseID: 500457). The project is assessed by the Center for Information Security and Privacy in Research (SIKT), and the Privacy Commissioner at UiT The Arctic University of Norway regarding Data Protection Impact Assessment (DPIA). Initiation of the study will be pending upon approval by all parties.

ELIGIBILITY:
Inclusion Criteria:

* Patients who, after clinical examination at University hospital of Northern Norway (UNN) fill the criteria for a chronic non-malignant pain diagnosis according to ICD-10.
* Satisfy criteria for a comorbid insomnia
* Both first-time referrals and former referred patients.

Exclusion Criteria:

* A comorbid drug abuse diagnosis (ICD-10)
* An ongoing compensation and/or insurance case related to a health issue, illness or treatment
* Drug treatment using >100 morphine equivalents
* Participation in other group-based treatments at the UNN Pain Department or the Physical Outpatient Medical Clinic (must be completed before inclusion)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Insomnia symptoms | Baseline and post-test (3 months), plus follow-up at 3 and 12 months.
  The Bergen Insomnia Scale (5 items, item score range 0-7 days) assesses the number of days per week with nighttime sleeping symptoms lasting more than 30 minutes (SOL-sleep onset latency, WASO-wake after sleep onset and EMA-early morning awakening without regaining sleep), and daytime problems (in number of days per week) related to general dissatisfaction and functional problems in school, work or social life. Symptoms that have a duration of >3 months and occur more than >3 days a week satisfy the inclusion criteria for insomnia.
Insomnia diagnosis | Baseline and post-test (3 months)
  The Duke Structured Diagnostic Interview for Sleep Disorders (Norwegian version translated by National Competence Center of Sleep Medicine in Bergen). is used to determine whether the DSM-5 criteria for insomnia are met. It is also used to make a clinical judgement of whether patients having other sleep issues, such as restless legs or sleep apnea, should be excluded.
Actigraphy insomnia indicators (SOL, WASO and EMA in minutes) | Baseline and post-test (3 months), plus follow-up at 3 and 12 months.
  Actiwatch Spectrum Plus from Phillips Respironics is used to record motion and bright light exposure during sleep. The actigraphy clock is worn on the left arm for 7 days. Outcome variables are Sleep Onset Latency (SOL; duration in minutes from initiation to falling asleep), Wake After Sleep Onset (WASO; duration in minutes of nightly awakenings), and Early Morning Awakening (EMA; duration in minutes from last wakeup to leaving bed).
Actigraphy insomnia indicators (SE %) | Baseline and post-test (3 months), plus follow-up at 3 and 12 months.
  Actiwatch Spectrum Plus from Phillips Respironics is used to record motion and bright light exposure during sleep. The actigraphy clock is worn on the left arm for 7 days. Outcome variable is Sleep Efficiency (SE; proportion of sleeping time to total time spent in bed). SE% = Duration of time in sleep / Duration of time in bed.
Sleep diary insomnia indicators (SOL, WASO and EMA in minutes) | Between baseline and post-test (3 months): Five repeated measures across five weeks
  Subjects complete a sleep diary log for a week following their participation in each sleep intervention module. The weekly sleep log is used to find and adjust the recommended bedtime concerning the participant's sleep restriction schedule. But as a primary outcome, it estimates Sleep Onset Latency (SOL; duration in minutes from initiation to falling asleep), Wake After Sleep Onset (WASO; duration in minutes of nightly awakenings) and Early Morning Awakening (EMA; duration in minutes from last wakeup to leaving bed) as indicators of insomnia.

SECONDARY OUTCOMES:
Sleep brain activity as measured by a simplified polysomnography device, i.e., a Home Sleep Test (HST) | Baseline and post-test (3 months)
  The HST recordings provide a good picture of sleep architecture (duration and distribution of N1, N2, N3 and REM sleep). These recordings are made a minimum of two nights per patient, excluding the first night due to habituation effects on the following night. In addition, the arousal index is used to indicate sleep disturbances during the night. A HST device manufatured by Somnomedics GmbH is considered used.
Anxiety and depression (HADS) | Baseline and post-test (3 months), plus follow-up at 3 and 12 months
  The Hospital Anxiety and Depression Scale (HADS: 7 anxiety + 7 depression items) is scored separately for anxiety and depression (sum score range 0-21, higher scores represents worse symptoms). The HADS subscale scores indicates the level of non-vegetative symptoms of anxiety and depression. A much-used cut-off score ≥ 8 may be used as a diagnostic marker of anxiety or depression.
Quality of Life (EQ-5Q-5L) | Baseline and post-test (3 months), plus follow-up at 3 and 12 months
  The EQ-5Q-5L (5 items) is a broad self-reported quality of life index evaluating 5 dimensions (severity rating: 1-no problems, 5-extreme problems): mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. It additionally includes a single-item for general evaluation of overall health status using a visual analogue scale ranging from 0-worst possible health to 100-best possible health.
Fatigue (Chalder Fatigue Scale) | Baseline and post-test (3 months), plus follow-up at 3 and 12 months
  The Chalder Fatigue Scale (13 items) quantifies the degree of physical and mental exhaustion with 7 and 4 items, respectively. Items are scored from 0-problem present less often than usual to 3-problem present much more often than usual.
Pain intensity, interference and locations (BPI) | Baseline and post-test (3 months), plus follow-up at 3 and 12 months
  The Brief Pain Inventory (BPI) indexes pain intensity (4 items) and interference (7 items), as well as body localizations. The severity and interference scores range from 0-no pain to 10-pain as bad as you can imagine. Bodily locations of pain symptoms (no or yes) are indicated on a body map, which is summed.
Tolerance and Acceptance of chronic pain (CPAQ-R) | Baseline and post-test (3 months), plus follow-up at 3 and 12 months
  The Chronic Pain Acceptance Questionnaire (CPAQ-revised: 20 items) measures pain tolerance and acceptance. Items are scored 0-not true to 6-always true with higher scores reflecting more tolerance or acceptance.

OTHER OUTCOMES:
Mediator: Sleep hygiene (SHI) | Baseline and post-test (3 months), plus follow-up at 3 and 12 months
  The Sleep Hygiene Index (SHI) consist of 13 items scored from 0-always to 4-never. Higher scores reflect better sleep hygiene practices, such as less daytime napping, regular bedtime routines and awaits goin to bed until feeling calm and tired.
Hyperactivity (HAS) | Baseline and post-test (3 months), plus follow-up at 3 and 12 months
  The HAS (26 items) evaluates the inclination to introspect, think about feelings, respond intensely to unexpected stimuli, and behaviors in general that evoke cortical arousal. Participants rate how much they agree on a scale from 0-not at all to 3-extremely. High scores reflect increased general cerebral responsiveness.
Mediator: Dysfunctional beliefs and attitudes about sleep (DBAS) | Baseline and post-test (3 months), plus follow-up at 3 and 12 months
  The DBAS contains 16 items probing for attitudes on a scale ranging from 0-disagree strongly to 10-agree strongly. Higher scores reflect more rigid beliefs or attitudes towards the minimum need sleep or quality of sleep.
Mediator: Metacognitions about insomnia (MCQ-i) | Baseline and post-test (3 months), plus follow-up at 3 and 12 months
  The MCQ-i uses a short version including 15 items that are scored on a 4-point Likert scale (1-do not agree to 4-agree very much). Higher scores reflect stronger unhelpful metacognitive beliefs about sleep, such as "I must control bodily physical sensation before falling asleep".
Mediator: Insomnia catastrophizing Scale (ISC) | Baseline and post-test (3 months), plus follow-up at 3 and 12 months
  The ISC includes 20 items that participants rate on a 6-point scale (0-never to 5-always). Higher scores reflect a higher degree of cognitive catastrophizing, e.g., negative expectations for the night's sleep, or adverse health health consequences of sleeping too poorly.
Mediator: Pain Catastrophizing Scale (PCS) | Baseline and post-test (3 months), plus follow-up at 3 and 12 months
  The PCS covers 13 items assessing the inclination to catastrophize about having persistent pain and the potential for further adverse health effects. Items are rated from 0-not at all to 4-all the time with higher scores reflecting worse tendency for catastrophizing.

CONTACTS AND LOCATIONS:
Overall Officials: Oddgeir Friborg, PhD, Principal Investigator — UiT The Arctic University of Norway
Locations (1):
- UiT The Arctic University of Norway, Tromsø, Troms County, Norway

IPD SHARING:
Plan to Share IPD: No
The project will collect considerable information about the health and clinical status of the patients, and their clinical response. After the publication of the primary outcome results, we plan to conduct numerous additional secondary outcome and exploratory analyses (e.g., mediation and moderation effects). The timeline for the entire publication process is uncertain, and we prefer not to upload anonymized patient data until most of these data have been analyzed and published. However, researchers interested in reanalyzing published data may contact the principal investigator and apply for data access.

REFERENCES:
- [Derived] Rosenvinge JH, Bergvik S, Abeler K, Tvedt K, Berge T, Lang N, Wilhelmsen M, Danielsson L, Pettersen G, Friborg O. The "SleepWell" intervention for patients with insomnia and persistent pain: a study protocol for a randomised waiting-list controlled trial of a cognitive behavioural group therapy programme. Trials. 2025 Aug 27;26(1):314. doi: 10.1186/s13063-025-09041-z. PMID 40866978